CLINICAL TRIAL: NCT05374031
Title: The Multiple Sclerosis Intimacy and Sexuality Questionnaire-15 (MSISQ-15): Validation of the Turkish Version in Patients With Multiple Sclerosis
Brief Title: Multiple Sclerosis Intimacy and Sexuality Questionnaire
Status: Completed | Type: Observational
Sponsor: Bozok University (Other)
Responsible Party: Principal Investigator, hanife dogan, Assistant Professor, Bozok University
Other Study IDs: 2017-KAEK 189
Record Dates: First submitted 2022-05-02; First posted 2022-05-13 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Multiple Sclerosis; Sexual Dysfunction; Questionnaires
Keywords: Multiple sclerosis; questionnaires; sexual dysfunction; self-report
MeSH Terms: conditions — Multiple Sclerosis; Sexual Dysfunction, Physiological

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: descriptive study — descriptive study

SUMMARY:
Aims: This study aimed to psychometrically evaluate the Turkish version of the Multiple Sclerosis Intimacy and Sexuality Questionnaire (MSISQ-15) in women with MS.

Methods: The study included 130 women with MS. The Turkish linguistic validation process of the original English MSISQ-15 was performed according to standardized guidelines. Reliability analysis was evaluated with test-retest analysis and intra-class correlation (ICC). Internal consistency between the items was analyzed using the Cronbach's alpha coefficient. Item analysis results were used to assess the contribution of the items to the scale. In evaluating the validity of the scale, the relationship between the MSISQ and the Female Sexual Function Index (FSFI), the Multiple Sclerosis Quality of Life Questionnaire-54 (MSQOL-54), and the Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PSIQ-12) was investigated. Psychometric properties were analyzed using internal consistency, test-rest reliability, construct validity, and floor-ceiling effect.

ELIGIBILITY:
Inclusion Criteria:

* Women over the age of 18 who were literate,
* who did not have any mental problems preventing cooperation and understanding,
* who were diagnosed with MS

Exclusion Criteria:

* Having pelvic organ prolapse stage 2 or more;
* having a history of relapse in the past 30 days;
* experiencing loss of balance or gait disturbance caused by a condition other than MS;
* being pregnant; having a history of gynecological, urological and/or neurological surgery;
* having a history of cesarean or vaginal birth in the past six months;
* being sexually inactive; and, having urinary tract infections

Ages: 19 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Multiple Sclerosis women
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2021-08-12 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2022-03-10 (Actual)

PRIMARY OUTCOMES:
Questionnaire | day 1
  Multiple Sclerosis Intimacy and Sexuality Scale is a 15-item self-report measure that assesses the impact of MS symptoms on sexual activity and satisfaction over the past 6 months.Higher scores indicate greater sexual problems.
Questionnaire | day 1
  Female Sexual Function Index is a 19-item scale that evaluates the sexual functions of female patients. The questionnaire consists of 6 separate subdimensions: desire, arousal, lubrication, orgasm, satisfaction, and pain. Higher scores indicate better sexual function.
Questionnaire | day 1
  Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire is an instrument that evaluates sexual function in women with urinary incontinence and/or pelvic organ prolapse. Increasing scores indicate better sexual function.
Questionnaire | day 1
  Global Pelvic Floor Bother Questionnaire is used to evaluate the presence and severity of the most common clinical problems caused by the pelvic floor dysfunction, namely, stress urinary incontinence, frequent and sudden urination sensation, urge incontinence, voiding difficulty, pelvic organ prolapse, obstructive defecation, fecal incontinence, and dyspareunia. A high score indicates more pelvic floor symptom complaints.
Questionnaire | day 1
  Multiple Sclerosis Quality of Life Questionnaire-54 is used to evaluate the quality of life of patients with MS. Higher scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Yozgat Bozok University, Yozgat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided